CLINICAL TRIAL: NCT07067112
Title: Suppressive Functions of Regulatory T Cells in Migraine
Acronym: SIIM-reg
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2025 MOISSET
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-06

CONDITIONS: Chronic Migraine
Keywords: Migraine; Inflammation; Immune system; Regulatory T cells
MeSH Terms: conditions — Migraine Disorders; Inflammation | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in either the chronic migraine or control group for comparison between chronic migraine patients and controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic migraine (Experimental): Chronic migraine patients will donate 100 milliliters (mL) of peripheral and venous blood, answer a questionnaire and 2 phone calls (one at day 1 and the other at day 3 from the blood test).
  Interventions: Biological: Blood sampling, questionnaire and phone call
- Controls (Experimental): Non-migraine controls will donate 100 mL of peripheral and venous blood, answer a questionnaire and 2 phone calls (one at day 1 and the other at day 3 from the blood test).
  Interventions: Biological: Blood sampling, questionnaire and phone call

INTERVENTIONS:
Biological: Blood sampling, questionnaire and phone call — The blood sample will drawn after a fasting period of at least 8 hours, and the questionnaire will be auto-administered

SUMMARY:
Migraine is a frequent, disabling condition, of great social and economical impact worldwide. This condition is more frequent in women and subjects with autoimmune and/or inflammatory diseases. Cytokine and immune cell dysregulations have been evidenced in migraine. Inflammation seems to play an important role in migraine chronification; however, the inflammatory mechanisms involved in migraine pathophysiology remain unclear. Regulatory T (Treg) cells play a central role in maintaining immune homeostasis. They regulate effector T (Teff) cell proliferation and cytokine production, through several suppressive mechanisms, such as the hydrolysis of adenosine triphosphate (ATP) into adenosine (ADO), mediated by surface enzymes Cluster Differentiation 39 (CD39) and Cluster Differentiation 73 (CD73). ATP is involved in pain processes in migraine, and insufficient hydrolysis could participate in pain chronification. Recent studies suggest altered proportions of Treg cells in migraine, and decreased levels of CD39-positive (CD39+) Treg cells, suggesting Treg suppressive functions may be decreased in the disease. However, there have been no functional studies to date to confirm this hypothesis.

The investigators believe Treg suppressive functions may be decreased in migraine, and that such alterations may be caused by a malfunction in the ADO pathway.

DETAILED DESCRIPTION:
Migraine is a major and global public health concern that affects 14% of the population worldwide. It is 2 to 3 times more prevalent in women than men and is the second leading cause of disability. Many patients remain unresponsive to currently available treatments. As evidenced in different studies, including our own, several auto-immune and inflammatory disorders, such as multiple sclerosis, are associated with a higher prevalence of migraine and a higher risk for migraine chronification (at least 15 headache days per month) compared to the general population. These findings suggest that inflammation may play an important role in migraine chronification. Cytokine and immune cell dysregulations have been evidenced in the disease but the role of inflammation in migraine pathophysiology remains unclear. Among T lymphocytes, regulatory T (Treg) cells play an important role in maintaining immune homeostasis. They regulate pro-inflammatory effector T (Teff) cells and proinflammatory cytokine release (IL-6, IL-17, interferon-γ) through different suppressive mechanisms such as the hydrolysis of pro-inflammatory and nociceptive adenosine triphosphate (ATP) into anti-inflammatory and antinociceptive adenosine (ADO), by Treg surface enzymes CD39 and CD73, present on 40% and 6-10% of Treg cells, respectively. ADO then suppresses Teff cells by binding to their ADO receptor A2A. ATP is involved in the transduction of pain signals in migraine and its insufficient hydrolysis can lead to pain chronification. It has been evidenced that Tregs naturally suppress interferon (IFN)-γ production by Teff cells. Their CD39-positive (CD39+) subsets also suppress IL-17 production by Teff cells, whereas CD39-negative (CD39-) Tregs seem to increase IL-17 secretion. Recent studies have shown altered Treg proportions in migraine compared to controls and Treg subpopulation dysregulations, such as decreased CD39+Treg cell levels. This further suggests that Treg suppressive functions may be altered in migraine, but no functional assays have been led to confirm that.

In this study, the investigators aim to determine whether Treg cells play a role in migraine pathophysiology, by answering the following 3 separate questions: Question 1) Are Treg suppressive functions decreased in migraine patients? Question 2) Are CD39+Treg cells functionally deficient in migraine patients? Question 3) Is the hydrolytic activity of enzyme CD39 reduced in migraine patients?

Through Treg/Teff coculture the investigators will assess the ability of total Treg and CD39+Treg cells to inhibit Teff proliferation and pro-inflammatory cytokine secretion and measure the hydrolytic activity of Treg enzyme CD39 on ATP in chronic migraine patients versus healthy controls. The use of human immune cells (Treg and Teff lymphocytes) in our experiments will allow the investigators to better understand migraine pathophysiology, with a direct application to human subjects, as well as to avoid animal testing and suffering. Through its animal-free setting, following the 'Reduce, Refine, Replace (3Rs)' principle, the investigators wish to promote animal-free research and the reduction of animal use for reagent production by using recombinant antibodies for flow cytometry and synthetic medium supplements for cell culture. This study will lead to a better understanding of the role of inflammation and Treg cells in migraine pathophysiology and will provide new perspectives for the development of personalized treatments according to the immune pain profile of migraine patients.

The investigators aim to show that Treg suppressive functions are altered in migraine and that the ADO pathway is deficient. Through Treg/Teff coculture the investigators will measure the ability of Tregs to inhibit Teff proliferation and cytokine secretion and assess the CD39-related hydrolytic activity of Tregs. This will allow the investigators to study Treg cells suppressive functions on Teff cells in female patients with chronic migraine and healthy female control participants.

ELIGIBILITY:
Inclusion Criteria:

* Females
* 18 to 50 years old
* Chronic migraine participants : chronic migraine (at least 15 days of headache/month, according to the International Classification of Headache Disorders, 3rd edition criteria

Exclusion Criteria:

* BMI < or = 17kg/m² or > or = 30kg/m²
* Diagnosis or suspicion of type 2 diabetes, auto-immune or inflammatory diseases, immunodeficiency diseases
* Diagnosis of headache of non-migraine origin, except for tension type headache < or = 4 days per month (i.e.: cluster headache, post-traumatic headache, cerebral tumour…)
* Pregnancy, delivery, miscarriage, breastfeeding, participation in a medically assisted human reproduction program (ovary stimulation/hormone therapy) < 3 months before blood sampling
* Menopause, hysterectomy, or bilateral oophorectomy
* Flare of the autoimmune/inflammatory disease of interest < 1 month before blood sampling
* Modification of maintenance therapy for the autoimmune/inflammatory disease of interest (start, change of molecule, interruption) < 3 months before blood sampling
* Modification of prophylactic anti-migraine therapy (start, change of molecule, interruption) < 3 months before blood sampling (for migraine participants)
* Hormone therapy (besides contraception and treatment of endometriosis)
* Transplantation (solid organ or bone marrow)
* Cancer (active or remitting) < 1 year before blood sampling (solid organ or blood)
* Haematologic disease (benign or malignant) of the lymphoid lineage
* Guardianship, curatorship, safeguard of justice or deprivation of liberty
* For controls : diagnosis of migraine

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Treg cell suppressive functions | Day 0
  To measure the suppressive effect of Treg cells on Teff cells in chronic migraine patients and healthy controls

SECONDARY OUTCOMES:
CD39+ Treg cell suppressive functions | Day 0
  To measure the suppressive effect of CD39+Treg cells on Teff cells in chronic migraine patients and healthy controls
CD39 activity | Day 0
  To measure the hydrolytic activity of Treg enzyme CD39 in chronic migraine patients and healthy controls
Cytokines | Day 0
  To measure the levels of cytokine levels in blood : interleukin (IL)-6, IL-10, IL-17, IFN-g and transforming growth factor b

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MOISSET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stovner LJ, Hagen K, Linde M, Steiner TJ. The global prevalence of headache: an update, with analysis of the influences of methodological factors on prevalence estimates. J Headache Pain. 2022 Apr 12;23(1):34. doi: 10.1186/s10194-022-01402-2. PMID 35410119
- [Background] Ashina M. Migraine. N Engl J Med. 2020 Nov 5;383(19):1866-1876. doi: 10.1056/NEJMra1915327. No abstract available. PMID 33211930
- [Background] Barbanti P, Aurilia C, Egeo G, Torelli P, Proietti S, Cevoli S, Bonassi S; Italian Migraine Registry study group. Late Response to Anti-CGRP Monoclonal Antibodies in Migraine: A Multicenter Prospective Observational Study. Neurology. 2023 Sep 12;101(11):482-488. doi: 10.1212/WNL.0000000000207292. Epub 2023 Apr 18. PMID 37072224
- [Background] Moisset X, Giraud P, Dallel R. Migraine in multiple sclerosis and other chronic inflammatory diseases. Rev Neurol (Paris). 2021 Sep;177(7):816-820. doi: 10.1016/j.neurol.2021.07.005. Epub 2021 Jul 27. PMID 34325914
- [Background] Moisset X, Ouchchane L, Guy N, Bayle DJ, Dallel R, Clavelou P. Migraine headaches and pain with neuropathic characteristics: comorbid conditions in patients with multiple sclerosis. Pain. 2013 Dec;154(12):2691-2699. doi: 10.1016/j.pain.2013.07.050. Epub 2013 Aug 2. PMID 23911697
- [Background] Edvinsson L, Haanes KA, Warfvinge K. Does inflammation have a role in migraine? Nat Rev Neurol. 2019 Aug;15(8):483-490. doi: 10.1038/s41582-019-0216-y. Epub 2019 Jul 1. PMID 31263254
- [Background] Thuraiaiyah J, Erritzoe-Jervild M, Al-Khazali HM, Schytz HW, Younis S. The role of cytokines in migraine: A systematic review. Cephalalgia. 2022 Dec;42(14):1565-1588. doi: 10.1177/03331024221118924. Epub 2022 Aug 12. PMID 35962530
- [Background] Nurkhametova D, Kudryavtsev I, Khayrutdinova O, Serebryakova M, Altunbaev R, Malm T, Giniatullin R. Purinergic Profiling of Regulatory T-cells in Patients With Episodic Migraine. Front Cell Neurosci. 2018 Sep 25;12:326. doi: 10.3389/fncel.2018.00326. eCollection 2018. PMID 30319363
- [Background] Loza MJ, Anderson AS, O'Rourke KS, Wood J, Khan IU. T-cell specific defect in expression of the NTPDase CD39 as a biomarker for lupus. Cell Immunol. 2011;271(1):110-7. doi: 10.1016/j.cellimm.2011.06.010. Epub 2011 Jul 18. PMID 21763644
- [Background] Vignali DA, Collison LW, Workman CJ. How regulatory T cells work. Nat Rev Immunol. 2008 Jul;8(7):523-32. doi: 10.1038/nri2343. PMID 18566595
- [Background] Giniatullin R, Nistri A, Fabbretti E. Molecular mechanisms of sensitization of pain-transducing P2X3 receptors by the migraine mediators CGRP and NGF. Mol Neurobiol. 2008 Feb;37(1):83-90. doi: 10.1007/s12035-008-8020-5. Epub 2008 May 6. PMID 18459072
- [Background] Fletcher JM, Lonergan R, Costelloe L, Kinsella K, Moran B, O'Farrelly C, Tubridy N, Mills KH. CD39+Foxp3+ regulatory T Cells suppress pathogenic Th17 cells and are impaired in multiple sclerosis. J Immunol. 2009 Dec 1;183(11):7602-10. doi: 10.4049/jimmunol.0901881. Epub 2009 Nov 16. PMID 19917691
- [Background] Faraji F, Shojapour M, Farahani I, Ganji A, Mosayebi G. Reduced regulatory T lymphocytes in migraine patients. Neurol Res. 2021 Aug;43(8):677-682. doi: 10.1080/01616412.2021.1915077. Epub 2021 Apr 14. PMID 33853506
- [Background] Arumugam M, Parthasarathy V. Reduction of CD4(+)CD25(+) regulatory T-cells in migraine: Is migraine an autoimmune disorder? J Neuroimmunol. 2016 Jan 15;290:54-9. doi: 10.1016/j.jneuroim.2015.11.015. Epub 2015 Nov 28. PMID 26711570
- [Background] Yang L, Zhou Y, Zhang L, Wang Y, Zhang Y, Xiao Z. Aryl hydrocarbon receptors improve migraine-like pain behaviors in rats through the regulation of regulatory T cell/T-helper 17 cell-related homeostasis. Headache. 2023 Sep;63(8):1045-1060. doi: 10.1111/head.14599. Epub 2023 Aug 4. PMID 37539825
- [Background] Anaya JM. Common mechanisms of autoimmune diseases (the autoimmune tautology). Autoimmun Rev. 2012 Sep;11(11):781-4. doi: 10.1016/j.autrev.2012.02.002. Epub 2012 Feb 12. PMID 22353402
- [Background] Guo Z, Zhang J, Liu X, Unsinger J, Hotchkiss RS, Cao YQ. Low-dose interleukin-2 reverses chronic migraine-related sensitizations through peripheral interleukin-10 and transforming growth factor beta-1 signaling. Neurobiol Pain. 2022 Jun 13;12:100096. doi: 10.1016/j.ynpai.2022.100096. eCollection 2022 Aug-Dec. PMID 35733705
- [Background] Okimura H, Tanaka Y, Fujii M, Shimura K, Maeda E, Ito F, Khan KN, Nakamura Y, Mori T, Kitawaki J. Changes in the proportion of regulatory T cell subpopulations during menstrual cycle and early pregnancy. Am J Reprod Immunol. 2022 Dec;88(6):e13636. doi: 10.1111/aji.13636. Epub 2022 Oct 21. PMID 36217280
- [Background] Douge A, Vituret C, Carraro V, Parry L, Coudy-Gandilhon C, Lemal R, Combaret L, Maurin AC, Averous J, Jousse C, Bay JO, Verrelle P, Fafournoux P, Bruhat A, Rouzaire P. Temporal regulation of transgene expression controlled by amino acid availability in human T cells. HLA. 2024 Jan;103(1):e15252. doi: 10.1111/tan.15252. Epub 2023 Oct 17. PMID 37848366